CLINICAL TRIAL: NCT07011693
Title: Switching Medication and Augmentation Strategies for SSRI-Resistant Adolescent Depression（SMART-I): An Open-Label, Multicenter, Randomized Controlled Trial
Brief Title: Switching Medication and Augmentation Strategies for SSRI-Resistant Adolescent Depression（SMART-I)
Acronym: SMART-I
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xinyu Zhou (Other)
Responsible Party: Sponsor-Investigator, Xinyu Zhou, Professer, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1stChongqingCQMU
Record Dates: First submitted 2025-05-26; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: adolescent; SSRI; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Sertraline; agomelatine; Aripiprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1-sertraline (Experimental): dosage form: po dosage:25-200mg frequency:qd duration: patients will be given sertraline as a switching treatment to SSRI.
  Interventions: Drug: Sertraline
- Group 2-agomelatine (Experimental): dosage form: po dosage:25-50mg frequency:qd duration: patients will be given agomelatine as a switching treatment to SSRI.
  Interventions: Drug: Agomelatine
- Group 3-aripiprazole with original SSRI (Experimental): dosage form: po dosage: 1.25-15mg frequency:qn duration: patientswill be given aripiprazole as an add-on treatment to original SSRI.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Sertraline — Commonly used oral antipsychotics intervention therapy.
  Arms: Group1-sertraline
Drug: Agomelatine — Commonly used oral antipsychotics intervention therapy.
  Arms: Group 2-agomelatine
Drug: Aripiprazole — Commonly used oral antipsychotics intervention therapy.
  Arms: Group 3-aripiprazole with original SSRI

SUMMARY:
This project aims to investigate the effectiveness of existing common antidepressants in adolescents with MDD who did not respond to their first treatment.

DETAILED DESCRIPTION:
This project aims to investigate the effectiveness of existing common antidepressants in adolescents with MDD who did not respond to their first treatment. Adolescents ages 12 to 17, currently taking a prescribed selective serotonin reuptake inhibitor (SSRI) at least 8 weeks and still experiencing depression, participate in a 8-week randomized treatment study that includes one of three conditions: (1) switching to sertraline , (2) switching to duloxetine , (3) augmentation of their original SSRI with aripiprazole.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 12-17;
2. As assessed by K-SADS-PL, it meets the DSM-5 criteria for MDD;
3. CDRS-R≥45;
4. CGI-S≥4;
5. Failed to respond to an initial SSRI trial: the trial at least 8 weeks, with the last of which were at a dosage of at least 40 mg per day of fluoxetine or its equivalent.

Exclusion Criteria:

1. Current or lifetime diagnosis of bipolar disorder, schizophrenia, autism, attention-deficit/hyperactivity disorder or obsessive-compulsive disorder or psychosis not otherwise specified;
2. MDD with psychotic symptoms;
3. YMRS>13;
4. Current or lifetime diagnosis of serious neurologic diseases such as epilepsy, brain trauma or other serious physical illnesses;
5. Failure to respond adequately to two or more antidepressant treatment trials of recommended dose and length (at least 8 weeks, with the last 4 of which were at a dosage of at least 40 mg per day of fluoxetine or its equivalent);
6. History of clear-cut intolerability of, or lack of effect with, an adequate trial of sertraline, agomelatine, or aripiprazole;
7. Current depressive episode with clear suicidal plans or behaviors;
8. Received modified electroconvulsive therapy within 3 months;
9. Taking any medicine that contraindicates in combination with or interferes with the efficacy of the treatment;
10. Substance abuse or dependence;
11. Female patients with pregnancy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
response rate of Children's Depression Rating Scale (CDRS-R) scores | Baseline of treatment period, 4 weeks, 8 weeks
  The primary outcomes are the treatment response rate (reduction rate of CDRS-R≥50%). The CDRS-R is a scale consisting of 17 items that are evaluated by clinicians to assess the intensity of depressive symptoms in adolescents, with items scored on scales of 1 to 5 or 1 to 7, resulting in a possible total score range of 17 to 113，higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in Baker Depression Scale（BDI-II) scores from baseline | Baseline of treatment period, 4 weeks, 8 weeks
  Change in BDI-II scores from baseline，The BDI is a self-report rating scale containing 21 items. Based on the BDI scores, depression can be classified into six levels: normal (1-10), mild mood disorder (11-16), borderline clinical depression (17-20), moderate depression (21-30), severe depression (31-40), and extreme depression (over 40).Higher scores mean a worse outcome.
Change in The Screen for Child Anxiety-Related Emotional Disorders (SCARED) scores from baseline | Baseline of treatment period, 4 weeks，8 weeks
  The SCARED is employed to evaluate child anxiety symptoms. Each question is rated from 0 to 2, with 0 denoting "not true or hardly ever true," 1 denoting "somewhat true or sometimes true", and 2 denoting "extremely true or often true". The maximum total score is 63. Higher scores mean a better or worse outcome.
Change in CGI-S (Clinical Global Impressions-Severity Scales) scores from baseline | Baseline of treatment period, 4 weeks, 8 weeks,
  Improvement in overall clinical impression severity（ 7-point scale, with 1 being normal and 7 being among the most severely damaged
Adverse Event (AE) or Serious Adverse Event (SAE) | Baseline of treatment period, 1 month, 2 months,
  Change in suicide risk from baseline on the C-SSRS (Columbia Suicide Severity Rating Scale), Adverse Event (AE) or Serious Adverse Event (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China